CLINICAL TRIAL: NCT00973791
Title: Fluid Management for Cesarean Section Undergoing Spinal Anesthesia
Brief Title: Fluid Management for Cesarean Section II
Acronym: FMCS-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: Nanjing Maternity and Child Health Care Hospital (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NJMU-08711MZ
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Cesarean Section
Keywords: Spinal anesthesia; Fluid therapy
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Prior crystalloid (Active Comparator): Crystalloid (Ringer's Lactate) was given before spinal anesthesia
  Interventions: Drug: Ringer's Lactate
- Posterior crystalloid (Active Comparator): Crystalloid (Ringer's Lactate) was given after spinal anesthesia
  Interventions: Drug: Ringer's Lactate
- Prior colloid (Active Comparator): Colloid (6% hydroxyethyl starch) was given before spinal anesthesia
  Interventions: Drug: Six percent hydroxyethyl starch
- Posterior colloid (Active Comparator): Colloid (6% hydroxyethyl starch) was given after spinal anesthesia
  Interventions: Drug: Six percent hydroxyethyl starch

INTERVENTIONS:
Drug: Ringer's Lactate — Ringer's Lactate 8 ml/kg was given intravenously before or after spinal anesthesia in cesarean section
  Other Names: Lactated Ringer's solution
  Arms: Posterior crystalloid; Prior crystalloid
Drug: Six percent hydroxyethyl starch — Hydroxyethyl starch (6%) was given before or after spinal anesthesia in cesarean section
  Other Names: HES/HAES
  Arms: Posterior colloid; Prior colloid

SUMMARY:
Fluid management plays an essential role in cesarean section. In previous study (NCT00488111) the investigators found that prior-epidural anesthesia fluid management produced a more significant role in stabilizing the blood pressure and better prognosis after cesarean delivery than that of the posterior-anesthesia ones. Given epidural anesthesia has a time interval before reaching the best state of anesthesia, so the fluid management also has a relatively adequate time to resuscitation. In reality, spinal anesthesia is used popularly except for the epidural anesthesia, whereas spinal anesthesia would produce more significant fluctuation of the hemodynamics compared with the latter. Herein the investigators proposed whether the prior-spinal anesthesia fluid management also produced similar effect on hemodynamic characteristics to the epidural anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 21-40 yr
* First time of delivery
* ASA status I-II
* No premature
* No genetic and infectious diseases
* Chinese

Exclusion Criteria:

* < 21 yr
* > 40 yr
* Subjects with cardiac and pulmonary disorders
* Dislocation of placenta
* Pregnant hypertension
* Allergy to local anesthetics
* Unwilling to cooperation
* Need intraoperative administration of vascular active agents
* With significant delivery side effects

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 860 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Rate of hypotension | Anesthesia begin (0 min) to 120 min after anesthesia

SECONDARY OUTCOMES:
Recurrence of hypotension after ephedrine or phenylephrine | Anesthesia begin (0 min) to 120 min after anesthesia
Consumption of ephedrine and phenylephrine | Anesthesia begin (0 min) to 120 min after anesthesia
Total volume of colloid or crystalloid | Fifteen minutes before anesthesia to 120 min after anesthesia
One-min and 5-min Apgar scores | The first and fifth minute after cesarean successful delivery
Oxygen saturation during hypotension | Anesthesia begin (0 min) to 120 min after anesthesia
Duration of hypotension | Anesthesia begin (0 min) to 120 min after anesthesia
Low umbilical cord pH (artery < 7.20) | At the time of successful delivery (0 min)

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- The Affiliated Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China